CLINICAL TRIAL: NCT03380767
Title: Use of Viscoelastic Tests in the Treatment of Trauma-induced Coagulopathy: a Pragmatic Randomized Clinical Trial Comparing Viscoelastic Tests With Conventional Assays.
Brief Title: Use of Viscoelastic Tests in the Treatment of Traumatic Induced Coagulopathy: a Pragmatic Randomized Clinical Trial.
Acronym: VISCOTRAUMA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Stefano Magnone, Attending General Surgeon, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trauma Study
Record Dates: First submitted 2017-12-17; First posted 2017-12-21 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Trauma, Multiple; Coagulopathy; Massive Hemorrhage
Keywords: trauma-induced coagulopathy
MeSH Terms: conditions — Multiple Trauma; Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POC group (Experimental): In this group, patients will be treated according to the information gathered by TEG or ROTEM assays.
  Interventions: Procedure: Trauma-induced coagulopathy treatment
- Conventional group (Experimental): In this group, patients will be treated according to the information gathered by conventional laboratory assays (platelet count, fibrinogen level, PT or INR and d dimer for fibrinolysis)
  Interventions: Procedure: Trauma-induced coagulopathy treatment

INTERVENTIONS:
Procedure: Trauma-induced coagulopathy treatment — Transfusion as needed according to the assay methodology

SUMMARY:
Trauma is the leading cause of death in young people. Trauma-induced coagulopathy (TIC) encompasses several aspects of traumatic bleeding. Monitoring of coagulopathy comprises use of Point-of-Care (POC) methods, such as thromboelastography (TEG) or Thromboelastometry (ROTEM) and conventional laboratory assays (platelet count, fibrinogen level, and PT or INR).

POC tests are thought to have a better performance on mortality and bleeding control than conventional tests. The aim of this study is to compare POC and conventional assays with plasma consumption as a primary outcome and 28 days mortality as a secondary one.

ELIGIBILITY:
Inclusion Criteria: all adult (> 18 years old) trauma patients treated in our Emergency Department with a TASH score > 18

Exclusion Criteria:

* dead on arrival
* no blood product administered after randomization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Fresh frozen plasma consumption | 3 years
  In the POC group plasma consumption is estimated 20% less than in conventional assays group

SECONDARY OUTCOMES:
Mortality | 28 days
  28 days mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Papa Giovanni XXIII, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez E, Moore EE, Moore HB. Management of Trauma-Induced Coagulopathy with Thrombelastography. Crit Care Clin. 2017 Jan;33(1):119-134. doi: 10.1016/j.ccc.2016.09.002. PMID 27894492
- [Background] Gonzalez E, Moore EE, Moore HB, Chapman MP, Chin TL, Ghasabyan A, Wohlauer MV, Barnett CC, Bensard DD, Biffl WL, Burlew CC, Johnson JL, Pieracci FM, Jurkovich GJ, Banerjee A, Silliman CC, Sauaia A. Goal-directed Hemostatic Resuscitation of Trauma-induced Coagulopathy: A Pragmatic Randomized Clinical Trial Comparing a Viscoelastic Assay to Conventional Coagulation Assays. Ann Surg. 2016 Jun;263(6):1051-9. doi: 10.1097/SLA.0000000000001608. PMID 26720428
- [Background] Hunt H, Stanworth S, Curry N, Woolley T, Cooper C, Ukoumunne O, Zhelev Z, Hyde C. Thromboelastography (TEG) and rotational thromboelastometry (ROTEM) for trauma induced coagulopathy in adult trauma patients with bleeding. Cochrane Database Syst Rev. 2015 Feb 16;2015(2):CD010438. doi: 10.1002/14651858.CD010438.pub2. PMID 25686465